CLINICAL TRIAL: NCT05241119
Title: Precise Treatment of Axillary Lymph Nodes After Neoadjuvant Chemotherapy Guided by Long-term Nanocarbon Tracing: a Clinical Cohort Study
Brief Title: Axillary Lymph Node Treatment Guided by Naocarbon Tracing After Neoadjuvant Chemotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Jianyi Li, Principal Investigator, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Shengjing-LJY06
Record Dates: First submitted 2021-12-21; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Breast Cancer
Keywords: Breast cancer, neoadjuvant chemotherapy, lymph nodes, nanocarbon
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SLNB Group (Experimental): undergo fluorescence SLNB
  Interventions: Procedure: SLNB
- pALND Group (Experimental): undergo low axillary lymph node dissection with ICBN as the boundary
  Interventions: Procedure: pALND
- ALND Group (Experimental): undergo ALND
  Interventions: Procedure: ALND

INTERVENTIONS:
Procedure: SLNB — undergo fluorescence SLNB.
  Arms: SLNB Group
Procedure: pALND — undergo low axillary lymph node dissection with ICBN as the boundary
  Arms: pALND Group
Procedure: ALND — undergo ALND
  Arms: ALND Group

SUMMARY:
For patients with early breast cancer with negative axillary lymph nodes, sentinel lymph node biopsy (SLNB) can largely avoid complications such as upper limb lymphoedema caused by axillary lymph node dissection (ALND). Locally advanced breast cancer requires neoadjuvant chemotherapy (NAC), based on the breast cancer treatment guidelines. In addition to shrinking the primary breast lesion, NAC can reduce the stage for axillary positive lymph nodes. Therefore, in recent years clinicians have been considering SLNB for patients whose axillary lymph nodes have turned negative after NAC. After verification by the clinical trials, the current NCCN guidelines recommend that patients with T1-3N0-1 undergo SLNB after NAC, however, the false negative rate (FNR) of conventional SLNB after NAC is as high as 14%, which potentially leads to underestimation of the risk for recurrence and metastasis, insufficient adjuvant therapy, eventually affects long-term survival. Thus, how to accurately assess and treat axillary lymph nodes after NAC remains an urgent clinical question to be answered.

In recent years, a method using a metal clip to label positive lymph node before NAC has emerged in order to reduce the FNR of SLNB after NAC. Its principle is to trace the metastasized lymph node, so that the lymph node can be accurately found in the surgery, even if the lymph node is not blue-stained at the time. Apparently, this method is more suitable for small number of nodes, and inappropriate for more than two metastasized nodes.

The diameter of manocarbon particles (150nm) is between that of lymphatic capillaries (120-500nm) and capillaries (20-50 nm). With the unique macrophage phagocytosis, nanocarbon particles can remain in the lymphatic system for a long time. Using nanocarbon to label positive lymph nodes before NAC, our pilot study explored the regression of axillary lymph nodes after NAC. We found that, except for a small number of drug-resistant patients, the regression of positive lymph nodes after NAC followed a pattern of from the superior to the inferior, and from the medial to the lateral. We also found that, the worse the efficacy of NAC, the fewer black-stained nodes after NAC, suggesting long-term tracing of positive axillary lymph nodes by nanocarbon particles can guide precise treatment of axillary lymph nodes after NAC. These findings are integrated with our previous research project which investigated the spatial distribution of positive axillary lymph nodes with the intercostals brachial nerve (ICBN) as the boundary. It is proposed that low lymph node dissection below ICBN (pALND) may be a safe and efficient method reducing lymphoedema in patients with negative nodes after NAC. Prone position CT scan combined with clinical palpation of axillary lymph nodes can comprehensively evaluate axillary conditions in patients with breast cancer before surgery, and determine node metastasis accurately, and make correct clinical plans.

DETAILED DESCRIPTION:
A total of 100 patients who are first diagnosed with breast cancer (stage N2 or N3) at the Liaoning Oncology Hospital will be recruited. Inclusive criteria: 1) Invasive breast cancer confirmed by biopsy and histology; 2) based on prone CT scan and Doppler ultrasound, axillary stage cN2-3; 3) agree and meet the requirements for NAC; 4) meet surgical requirements and agree to undergo surgery after NAC; 5) the regime of NAC follows the NCCN recommendations. Exclusive criteria: previous history of breast cancer or other malignant tumors. Period of investigation: 2 years.

After informed consent is obtained, under ultrasound guidance, the metastatic lymph node with the largest diameter (> 1 cm) is selected and injected under the cortex with 0.3 ml of nanocarbon. If the cortex and medulla are difficult to distinguish, inject on the surface of the node. Patients with efficacy for NAC should complete the scheduled cycles of NAC. Alteration of NAC regime is allowed for patients whose initial NAC is inefficacious, as guided by the physicians.

Surgery is performed within four weeks after completion of the last cycle of NAC. Axillary lymph nodes are assessed using CT scan. For patients with neoadjuvant efficacy of CR and PR, axillary surgery is performed under fluorescent tracing. SLNB is performed for patients with extensive black staining nodes. Standard ALND is performed if SLN is positive. For patients with less than three black-stained nodes, pALND will be performed rather than SLNB. If axilary lynph nodes under the ICBN are proved positive by frozen histology, ALND is then performed. For those with neoadjuvant efficacy of SD or PD, pALND will be performed if there are extensive black-stained nodes. Standard ALND will be performed if lymph nodes are positive as assessed by intraoperative frozen histology. ALND will be performed if the number of black-stained nodes is less than 3.

All the clinical information and imaging data will be securely preserved, including surgical procedure, black-stained and metastasized lymph nodes. Short-term observatory measures include axillary drainage (quantity, extubation time) and upper limb lymphatic drainage (changes in arm circumference 10cm above and below the elbow pre and post surgery. Long-term observatory measures include axillary recurrence rate and lymphoedema 3-5 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* invasive breast cancer confirmed by biopsy and histology;
* based on prone CT scan and Doppler ultrasound, axillary stage cN2-3;
* agree and meet the requirements for NAC;
* meet surgical requirements and agree to undergo surgery after NAC;
* the regime of NAC follows the NCCN recommendations.

Exclusion Criteria:

• previous history of breast cancer or other malignant tumors.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
post-surgery pathology concordance rate | up to 3 weeks
  post-surgery pathology concordance rate:investigate if the false negative rates in SLNB and ALND groups are consistent with post-surgery pathological results.

SECONDARY OUTCOMES:
Axillary drainage | up to 3 weeks
  daily quantity of drainage for patients
Upper limb lymphatic drainage | up to 5 years
  Upper limb lymphatic drainage:investigate the changes in aim circumference 10 cm above and below the elbow two weeks, six months, 12 months after surgery, among SLNB, pALND and ALND groups.
Axillary recurrence rate 3-5 years after surgery | up to 5 years
  Axillary recurrence rate 3-5 years after surgery:the time between the start of treatment and the first diagnosis of axillary recurrene.
Upper limb lymphoedema | up to 5 years
  Clinical judgment is mainly by asking the patient's subjective feelings or physical examination and performing a multi-segment ratio for measurement. It is generally determined that the peripheral diameter of the upper limb on the affected side is longer than the circumference of the contralateral upper limb< 3 cm is mild edema, 3 to 5 cm is moderate edema, and the > 5 cm is severe edema.

CONTACTS AND LOCATIONS:
Overall Officials: Jianyi Jianyi, Master, Principal Investigator — Cancer Hospital of China Medical University, Liaoning Cancer Hospital
Locations (2):
- China (2):
  - Cancer Hospital of China Medical University, Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - Jianyi Li, Shenyang, Liaoning